CLINICAL TRIAL: NCT02763007
Title: An Extension Study of Protocol ALO-IIT(PEAK Study) to Examine the Long-term Efficacy and Safety of Metformin + Alogliptin + Pioglitazone Triple Combination Therapy in the Korean Type 2 Diabetes Patients
Brief Title: An Extension Study of PEAK Trial
Acronym: PEAK-E
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty in recruiting patients
Sponsor: Kun-Ho Yoon (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Kun-Ho Yoon, professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEAK-E
Record Dates: First submitted 2016-04-29; First posted 2016-05-05 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- alogliptin+pioglitazone (Experimental): A group who treat with alogliptin+pioglitazone: The Combination of Alogliptin 25 mg and pioglitazone 30 mg daily add on metformin for 28 week as extension and followed by 2 years of observation
  Interventions: Drug: alogliptin+pioglitazone
- alogliptin (Active Comparator): A group who treat with alogliptin: Alogliptin 25 mg daily add on metformin for for 28 week as extension and followed by 2 years of observation
  Interventions: Drug: alogliptin
- pioglitazone (Active Comparator): A group who treat with pioglitazone: Pioglitazone 30 mg daily add on metformin for for 28 week as extension and followed by 2 years of observation
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: alogliptin+pioglitazone — alogliptin and pioglitazone add on metformin
  Other Names: nesina, actos
  Arms: alogliptin+pioglitazone
Drug: alogliptin — nesina add on metformin
  Other Names: nesina
  Arms: alogliptin
Drug: pioglitazone — actos add on metformin
  Other Names: actos
  Arms: pioglitazone

SUMMARY:
Double blind, three arm, comparative intervention trial for 24 weeks(PEAK study) with open label extension trial for 28 weeks followed by 2 year observational study.

DETAILED DESCRIPTION:
PEAK trial is now undergoing (Multicenter, randomized, double blind, three-arm parallel group study to evaluate efficacy and safety of Alogliptin and Pioglitazone combination therapy on glucose control in type 2 diabetes subjects who have inadequate control with Metformin monotherapy in Korea, Takeda No. ALO-IIT-012).

Duration of combination treatment is 24 week in the PEAK trial. Long-term efficacy and safety of alogliptin + pioglitazone + metformin combination therapy is not defined in Korea yet.

Thus, extension of the PEAK trial for the longer treatment upto 1 year has been planned.

PEAK trial will be followed by another 28 week open-label treatment of the same drug as initial randomization (total duration of treatment as randomized 52 week), and followed by 2 year of observation.

During observation period, any antidiabetic medication can be added/changed when HbA1c of the subject is off target 7% with clinician's clinical decision.

After 3 years of initial randomization, durability of glucose control will be assessed between 3 treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Completed "ALO-IIT-012(PEAK study)", without major protocol deviations.
* Male, or female, 19 years to 75 years.
* Female with childbearing potential who has a negative urine pregnancy test result at study start and willing to continue practice appropriate birth control during the entire duration of study
* Subjects completed PEAK can be included within 30 days after End Of the Study
* Subjects completed PEAK can be included if their treatment is the same as randomized even after 30 days of End Of the Study.

Exclusion Criteria:

* eGFR(Epidermal growth factor receptor) < 50mL/min
* AST(aspartate aminotransferase)/ALT(alanine aminotransaminase) >2.5 upper limit of normal
* Pregnant or lactating women
* Subject who the investigator deems inappropriate to participate in this study
* Patients with a history of bladder cancer or patients with active bladder cancer
* Patients with uninvestigated macroscopic hematuria
* Patients with cardiac failure or a history of cardiac failure (New York Heart Association [NYHA] Stages 3 to 4)
* Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, since this study drug contains lactose

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving HbA1c <7% after 36 month treatment | 36 months after randomization
  The proportion of subjects achieving HbA1c on target < 7.0% after 36 month.

SECONDARY OUTCOMES:
Proportion of subjects achieving HbA1c <6.5% after 36 month treatment | 36 Months after randomization
  The proportion of subjects achieving HbA1c on target < 6.5% after 36 month.
Proportion of subjects achieving HbA1c <7% after 12 month treatment | 12 Months after randomization
  The proportion of subjects achieving HbA1c on target < 7.0% after 12 month.
Change in glycated hemoglobin(HbA1c) from baseline to 12 month | baseline, 12 months
  Change from baseline in HbA1c after 6 month of double blinded treatment followed by 6 month open treatment
Change in HOMA-IR(homeostasis model assessment of insulin resistance) from baseline to 36 month | baseline, 36 months
  Change from baseline in HOMA-IR(homeostasis model assessment of insulin resistance) after 12 month of randomized treatment followed by 24 month observation.
change of HOMA-beta(homeostasis model assessment of beta cell) from baseline to 36 month | baseline, 36 months
  Change from baseline in HOMA-beta(homeostasis model assessment of beta cell) after 12 month of randomized treatment followed by 24 month observation.

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, MD, PhD, Principal Investigator — Seoul St Mary's Hospital, The Catholic University of Korea
Locations (1):
- Seoul St Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No